CLINICAL TRIAL: NCT04149886
Title: Cardiac Ganglionated Plexus Ablation Before Permanent Pacemaker Implantation in Patients With Sick Sinus Syndrome - A Multicenter, Randomized, Prospective Clinical Trial
Brief Title: Cardiac Ganglionated Plexus Ablation Before Permanent Pacemaker Implantation in Patients With Sick Sinus Syndrome
Acronym: GAPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: RenJi Hospital (Other); Heart Center of The First Affiliated Hospital of Xinjiang Medical Unviersity (Unknown); Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Yan Yao, MD,PhD, Chief of First Department of Arrythmia Center, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20191026
Record Dates: First submitted 2019-10-26; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Cardioneuroablation; Permanent Pacemaker Implantation; Sick Sinus Syndrome; Ganglionated Plexus
Keywords: Cardioneuromablation; Ganglionated plexus; Sick Sinus Syndrome; Pacing percentage
MeSH Terms: conditions — Sick Sinus Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ablation group(Ablation+pacemaker) (Experimental): The cardioneuroablation will be performed under conscious sedation. After 3-dimensional endocardial surface of the LA and pulmonary veins have been constructed by Ensite system, the GP sites can be located in LA；High frequecy stimulation（HFS）will be used to conform if there is a positive vagal response at each GP site. The upper limits of power and temperature will be set to 30-40 W and 43-60°C, respectively. And if no vagal response been induced during ablation, radiofrequency will be delivered for 30 seconds and stopped in this site. The end point of the ablation procedure will be that no vagal response could be induced by repeat HFS.
  After ablation of GPs, the participants will receive permanent pacemaker implantation(see arm of control group).
  Interventions: Procedure: cardiac ganglion plexus ablation(cardioneuroablation); Device: Permanent pacemaker implantation
- Control group(only pacemaker) (Sham Comparator): The control group only treated with permanent pacemaker without cardioneuroablation.The participants will receive permanent pacemaker implantation, the pacemaker placement will be done in accordance with standards at each center. All implanted pacemakers are provided two manufacturers (St. Jude Medical or Medtronics), His bundle pacing will be recommended in patients with a LVEF between 35%-45%. After placement of permanent pacemaker, the participants will be followed-up at 1 week, 3,6,12 months. After the permanent pacemaker implantation, the rate response function should be turned off and low pacing rate should be set at 60bpm uniformly in all the eligible participants.
  Interventions: Device: Permanent pacemaker implantation

INTERVENTIONS:
Procedure: cardiac ganglion plexus ablation(cardioneuroablation) — Cardiac ganglion plexus ablation in the left atrium will be performed before implanting permanent pacemaker in patients with sick sinus syndrome.
  Arms: Ablation group(Ablation+pacemaker)
Device: Permanent pacemaker implantation — DDD permanent pacemaker will be implanted in the paticipants.
  Other Names: St. Jude Medical or Medtronic

SUMMARY:
Different studies for cardiac ganglionated plexus（GP） ablation to treat vagal vascular syncope, sinus node dysfunction, and functional atrioventricular block have been published. Investigators have developed a more specific approach of cardiac, called cardioneuroablation . This treatment is based on a high-frequency stimulation (HFS) and/or anatomical landmarks to identify GPs in left atrium，which being targeted by radiofrequency catheter ablation. The feasibility of GPs ablation/cardioneuroablation has already been tested in our center in former studies in humans,with a favorable outcome for the patients involved. The results of the former studies have been submitted for publication. However, there are no prospective randomized studies to evaluate the efficacy and safety of atrial ganglionated plexus ablation for SSS before permanent pacemaker implantation.

The purpose of this study of GAPS in humans is to evaluate the efficacy and safety of cardioneuroablation in patients of sick sinus syndrome before they receive a permanent pacemaker.

DETAILED DESCRIPTION:
This is a multicenter,prospective, open, interventional study. All patients will undergo permanent pacemaker implantation. The study will involve eight different steps, from the screening procedure through study completion: screening, enrollment, pharmacological testing, randomization of group allocation, preprocedural assessment, procedure, follow-up, study completion. The dedicated study members (cardiac electrophysiologists, statisticians) and the PI are responsible for recording all data from the trial on the case report forms (CRFs) and completing the study database. The participants will be randomly allocated in a 1:1 ratio to either GPs ablation followed by permanent pacemaker implantation or pacemaker alone. Randomization will be conducted centrally by an independent statistics department(Oxford Medical Center of National Center for Cardiovascular Diseases, Beijing, China) and stratified by center and age(<50 or >=50 years); A dedicated independent physician will be responsible for the safety monitoring. The PI will permit inspection of the trial files and the database by national or international official controlling scientific authorities, if required. The PI will review and monitor completed CRFs and the database at regular intervals throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form.
* Diagnosed as SSS, with recurrent symptomatic bradycardia, blackouts, syncope, etc.
* Meet the indications for permanent pacemaker implantation according to the 2018 Chinese pacemaker guidelines (Class I, Class IIa).
* Positive reaction to atropine: The PP interval shortened by more than 20% or the sinus heart rate>60 bpm after intravenous injection of 2 mg of atropine.

Exclusion Criteria:

* Age <14 years old or >75 years old.
* Accompanied with complex congenital heart disease, valvular heart disease, cardiomyopathy and other chronic diseases, such as heart failure (NYHA grade III or IV).
* Acute coronary syndrome or myocardial infarction occurred within 6 months. Cerebrovascular events (such as transient ischemic attack, stroke) or other cerebral blood supply disorders occurred within 3 months.
* History of cardiac surgery and/or permanent cardiac pacemaker implantation.
* TEE or CT found a left atrial thrombus and/or left atrial anteroposterior diameter > 55mm or LVEF < 35%.
* Persistent atrial fibrillation, high-degree or complete atrioventricular block; double or triple fascicular block.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-28 (Estimated); Primary Completion 2020-10-27 (Estimated); Study Completion 2021-10-27 (Estimated)

PRIMARY OUTCOMES:
Percentage of atrial pacing of permanent pacemaker programming | 12 months （±14 days）
  Percentage of atrial pacing of permanent pacemaker at 12 months after the implantation of permanent pacemaker with program control.
Percentage of pacing of paced rhythm in Holter record | 1 week
  Percentage of pacing of paced rhythm in Holter record 1week after pacemaker implantation

SECONDARY OUTCOMES:
Percentage of sinus rhythm beats in Holter records | 1 week, 3 months(±5 days), 6 months (±7 days)，12 months （±14 days）
  Percentage of sinus rhythm beats at 1 week, 3 months, 6 months and 12 months with Holter.
Freedom from syncope | 1 week, 3 months(±5 days), 6 months (±7 days)，12 months （±14 days）
  Freedom from sycope at 1 week, 3 months, 6 months and 12 months with outpatient clinic follow up.
Improvement of quality of life: Short Form-36 (SF-36) or Euroqol (EQ-5D) | 1 week, 3 months(±5 days), 6 months (±7 days)，12 months （±14 days）
  Improvement of quality of life with questionair at 1 week, 3 months, 6 months and 12 months with outpatient clinic follow up.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - China National Center for Cardiovascular Diseases, Beijing, Beijing Municipality
  - 1Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qin M, Zhang Y, Liu X, Jiang WF, Wu SH, Po S. Atrial Ganglionated Plexus Modification: A Novel Approach to Treat Symptomatic Sinus Bradycardia. JACC Clin Electrophysiol. 2017 Sep;3(9):950-959. doi: 10.1016/j.jacep.2017.01.022. Epub 2017 Apr 26. PMID 29759719
- [Background] Debruyne P, Rossenbacker T, Collienne C, Roosen J, Ector B, Janssens L, Charlier F, Vankelecom B, Dewilde W, Wijns W. Unifocal Right-Sided Ablation Treatment for Neurally Mediated Syncope and Functional Sinus Node Dysfunction Under Computed Tomographic Guidance. Circ Arrhythm Electrophysiol. 2018 Sep;11(9):e006604. doi: 10.1161/CIRCEP.118.006604. PMID 30354289
- [Background] Cui B, Lu Z, He B, Hu X, Wu B, Xu S, Huang C, Jiang H. Acute effects of ganglionated plexi ablation on sinoatrial nodal and atrioventricular nodal functions. Auton Neurosci. 2011 Apr 26;161(1-2):87-94. doi: 10.1016/j.autneu.2011.01.004. PMID 21316313